CLINICAL TRIAL: NCT03233165
Title: Comparison Between Two Different High Power Ablative Lasers in the Treatment of Oral Leukoplakia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Dragana Gabrić, Clinical Professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-PA-26-6/2015
Record Dates: First submitted 2017-07-23; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Leukoplakic Lesions
Keywords: laser therapy; recurrence; leukoplakia; precancerous lesion
MeSH Terms: conditions — Leukoplakia; Recurrence | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with diagnosed leukoplakia 1 (Experimental): Patients who meet the conditions of pathohistological diagnosis of leukoplakia and clinical criteria for diagnosis of non-homogeneous leukoplakia.
  Intervention using Er:YAG laser
  Interventions: Procedure: Er:YAG laser
- Patients with diagnosed leukoplakia 2 (Experimental): Patients who meet the conditions of pathohistological diagnosis of leukoplakia and clinical criteria for diagnosis of non-homogeneous leukoplakia.
  Intervention using Er,Cr:YSGG laser
  Interventions: Procedure: Er,Cr:YSGG laser

INTERVENTIONS:
Procedure: Er:YAG laser — Ablation of the lesions Device: Er:YAG laser (LightWalker AT, Fotona, Slovenia, 2013) with a non-contact X-Runner digitally controled hand-piece.
  Settings for the Er:YAG laser were as follows: pulse mode was Quantum Square Pulse (QSP), pulse energy of 120mJ, frequency of 20Hz and water sprey level was set to10ml per minute.
  Arms: Patients with diagnosed leukoplakia 1
Procedure: Er,Cr:YSGG laser — Ablation of the lesions Device: Er,Cr:YSGG laser(WaterLase iPlus, Biolase LTD, USA) using contact mode. Settings were subsequent: power 50W, frequency 50Hz and concentration ratio of air and water was 2:4.
  Arms: Patients with diagnosed leukoplakia 2

SUMMARY:
Oral leukoplakia is a precancerous lesion with relatively high malignant transformation potential. They are often treated by wide surgical excisions or conservative retinoids therapy. The use of high power ablative lasers has been proposed as an effective way of treating these lesions safely. The aim of this study was to evaluate efficiency Er:YAG and Er,Cr:YSGG laser, in the treatment of oral leukoplakia.

DETAILED DESCRIPTION:
The purpose of this research was to determine the effectiveness of two high-power ablative lasers in the treatment of oral leukoplakia. Furthermore, the purpose was to compare reciprocally and evaluate the subjective and objective postoperative parameters for two different tested ablative lasers, Er: YAG and Er, Cr: YSGG.

All the patients were referred to the Department of Oral Medicine or Oral Surgery where a biopsy and measuring the size of lesion that meet the criteria of the histopathological diagnosis of leukoplakia was performed. Patients who met the conditions of pathohistological diagnosis of leukoplakia and clinical criteria for diagnosis of non-homogeneous leukoplakia, were included in the research.

The patients were randomly allocated into one of the two test groups. In the first group of patients leukoplakia lesion were removed using high-power ablative laser Er: YAG and to those in the second group using high power ablative Er, Cr: YSGG laser.

The patients were monitored one year and six months after treatment to evaluate subjective and objective parameters focused on life quality after treatment and in case of eventual relapse. Criteria of effectiveness for lasers were appearance of relaps in one year and six months following.

ELIGIBILITY:
Inclusion Criteria:

* based clinically diagnosed non homogeneous leukoplakia

Exclusion Criteria:

* immunocompromised patients
* HIV positive patients
* patients on suppressive therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 6 months period
  At a recall visit after six months there were no recurrence of all leukoplakia which were ablated by use of Er:YAG and Er;Cr:YSGG laser.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dragana Gabrić, Study Director — University of Zagreb

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Waal I, Schepman KP, van der Meij EH, Smeele LE. Oral leukoplakia: a clinicopathological review. Oral Oncol. 1997 Sep;33(5):291-301. doi: 10.1016/s1368-8375(97)00002-x. PMID 9415326
- [Background] Nair DR, Pruthy R, Pawar U, Chaturvedi P. Oral cancer: Premalignant conditions and screening--an update. J Cancer Res Ther. 2012 Jan;8 Suppl 1:S57-66. doi: 10.4103/0973-1482.92217. PMID 22322734
- [Background] van der Waal I, Axell T. Oral leukoplakia: a proposal for uniform reporting. Oral Oncol. 2002 Sep;38(6):521-6. doi: 10.1016/s1368-8375(01)00125-7. PMID 12167428
- [Background] Holmstrup P, Dabelsteen E. Oral leukoplakia-to treat or not to treat. Oral Dis. 2016 Sep;22(6):494-7. doi: 10.1111/odi.12443. Epub 2016 Feb 11. PMID 26785709
- [Background] van der Waal I. Potentially malignant disorders of the oral and oropharyngeal mucosa; present concepts of management. Oral Oncol. 2010 Jun;46(6):423-5. doi: 10.1016/j.oraloncology.2010.02.016. Epub 2010 Mar 21. PMID 20308005
- [Background] Azma E, Safavi N. Diode laser application in soft tissue oral surgery. J Lasers Med Sci. 2013 Fall;4(4):206-11. PMID 25606331
- [Background] Silverman S Jr, Gorsky M, Lozada F. Oral leukoplakia and malignant transformation. A follow-up study of 257 patients. Cancer. 1984 Feb 1;53(3):563-8. doi: 10.1002/1097-0142(19840201)53:33.0.co;2-f. PMID 6537892
- [Background] Montebugnoli L, Frini F, Gissi DB, Gabusi A, Cervellati F, Foschini MP, Marchetti C. Histological and immunohistochemical evaluation of new epithelium after removal of oral leukoplakia with Nd:YAG laser treatment. Lasers Med Sci. 2012 Jan;27(1):205-10. doi: 10.1007/s10103-011-0941-y. Epub 2011 Jun 18. PMID 21687980
- [Background] Lodi G, Porter S. Management of potentially malignant disorders: evidence and critique. J Oral Pathol Med. 2008 Feb;37(2):63-9. doi: 10.1111/j.1600-0714.2007.00575.x. PMID 18197849
- [Background] Schoelch ML, Sekandari N, Regezi JA, Silverman S Jr. Laser management of oral leukoplakias: a follow-up study of 70 patients. Laryngoscope. 1999 Jun;109(6):949-53. doi: 10.1097/00005537-199906000-00021. PMID 10369289
- [Background] Chu FW, Silverman S Jr, Dedo HH. CO2 laser treatment of oral leukoplakia. Laryngoscope. 1988 Feb;98(2):125-30. doi: 10.1288/00005537-198802000-00001. PMID 3123826
- [Background] White JM, Chaudhry SI, Kudler JJ, Sekandari N, Schoelch ML, Silverman S Jr. Nd:YAG and CO2 laser therapy of oral mucosal lesions. J Clin Laser Med Surg. 1998 Dec;16(6):299-304. doi: 10.1089/clm.1998.16.299. PMID 10204434
- [Background] Roodenburg JL, Panders AK, Vermey A. Carbon dioxide laser surgery of oral leukoplakia. Oral Surg Oral Med Oral Pathol. 1991 Jun;71(6):670-4. doi: 10.1016/0030-4220(91)90271-d. PMID 1905797
- [Background] Rossmann JA, Brown RS, Hays GL, Lusk SS. Carbon dioxide laser surgical therapy for the management of oral leukoplakia: a case report. Tex Dent J. 1994 Dec;111(12):17-9, 21. No abstract available. PMID 8633283
- [Background] Ishii J, Fujita K, Komori T. Laser surgery as a treatment for oral leukoplakia. Oral Oncol. 2003 Dec;39(8):759-69. doi: 10.1016/s1368-8375(03)00043-5. PMID 13679199
- [Background] Meister J, Franzen R, Eyrich G, Bongartz J, Gutknecht N, Hering P. First clinical application of a liquid-core light guide connected to an Er:YAG laser for oral treatment of leukoplakia. Lasers Med Sci. 2010 Sep;25(5):669-73. doi: 10.1007/s10103-010-0782-0. PMID 20393767
- [Background] Schwarz F, Maraki D, Yalcinkaya S, Bieling K, Bocking A, Becker J. Cytologic and DNA-cytometric follow-up of oral leukoplakia after CO2- and Er:YAG-laser assisted ablation: a pilot study. Lasers Surg Med. 2005 Jul;37(1):29-36. doi: 10.1002/lsm.20188. PMID 15954115
- [Background] Seoane J, Gonzalez-Mosquera A, Lopez-Nino J, Garcia-Caballero L, Aliste C, Seoane-Romero JM, Varela-Centelles P. Er,Cr:YSGG laser therapy for oral leukoplakia minimizes thermal artifacts on surgical margins: a pilot study. Lasers Med Sci. 2013 Nov;28(6):1591-7. doi: 10.1007/s10103-013-1266-9. Epub 2013 Jan 17. PMID 23324955